CLINICAL TRIAL: NCT05046639
Title: Sciatic Block in Contralateral Limb for Treatment of Refractory Phantom and Residual Limb Pain; a Triple-Blind Randomized Crossover Controlled Trial
Brief Title: Sciatic Block in Contralateral Limb Phantom and Residual Limb Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal investigator is leaving the university.
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00215101
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Pain; Amputation
Keywords: Pain; Amputation; Phantom Pain
MeSH Terms: conditions — Pain; Phantom Limb | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Crossover Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study pharmacy will prepare the study medication and it will be labeled as subject number for administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group 2% Lidocaine first, then Sham Preservative Free Saline (Experimental): Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
  Crossover: Image guided sciatic nerve anesthetic block of the contralateral limb with 10 mL preservative-free saline.
  Crossover treatment will occur 5 days after the first block.
  Interventions: Drug: 10 mL 2% lidocaine
- Sham Preservative Free Saline first, then Treatment Group 2% Lidocaine (Placebo Comparator): Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
  Crossover: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
  Crossover treatment will occur 5 days after the first block.
  Interventions: Drug: 10 mL preservative free saline

INTERVENTIONS:
Drug: 10 mL 2% lidocaine — Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine. Crossover treatment 5 days later using image guided sciatic nerve anesthetic block of the contralateral limb with 10 mL preservative-free saline.
  Arms: Treatment Group 2% Lidocaine first, then Sham Preservative Free Saline
Drug: 10 mL preservative free saline — Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
  Crossover treatment 5 days later using Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
  Arms: Sham Preservative Free Saline first, then Treatment Group 2% Lidocaine

SUMMARY:
Participants with chronic, refractory phantom limb pain (PLP) or residual limb pain (RLP) for more than 6 months will be enrolled in this clinical trial. Aim: Define the attributable pain relief and functional improvement in participants with PLP/RLP after contralateral limb sciatic nerve block. Also, contribute to the basic science understanding of the crossed-withdraw reflex by demonstrating a known animal model phenomenon in human participants. Hypothesis: Contralateral limb sciatic nerve anesthetic block with 2% lidocaine provides immediate clinically meaningful pain reduction, defined as the proportion of patients with at least 50% improvement in numeric rating scale (NRS) pain score in PLP/RLP when compared to sham.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age greater than 18 years of age at day of enrollment
* 2. Lower extremity amputation performed more than 12 months before study enrollment
* 3. PLP/RLP in affected amputated limb > 4 on numeric rating scale 26 (NRS26)
* 4. Pain duration of more than 6 months despite a trial of conservative therapies for at least 2 months, including oral medications, topical medicines, physical therapy, and physical modalities (i.e., heat, cold, transcutaneous electrical nerve stimulation, phonophoresis)
* 5. Willingness to undergo image guided diagnostic nerve block

Exclusion Criteria:

* 1. Refusal / inability to participate or provide consent
* 2. Contraindications to diagnostic nerve block
* 3. Non-neurogenic source of PLP/RLP
* 4. Current opioid use > 50 morphine milligram equivalents per day
* 5. Any interventional pain treatment in the residual limb within the last 30 days
* 6. Severe uncontrolled medical condition (i.e., hypertensive crisis, decompensated hypothyroidism)
* 7. Use of investigational pain drug within past 30 days or other concurrent clinical trial enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hogue, MD, Study Director — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richardson C, Glenn S, Horgan M, Nurmikko T. A prospective study of factors associated with the presence of phantom limb pain six months after major lower limb amputation in patients with peripheral vascular disease. J Pain. 2007 Oct;8(10):793-801. doi: 10.1016/j.jpain.2007.05.007. Epub 2007 Jul 12. PMID 17631056
- [Background] Cohen SP, Gilmore CA, Rauck RL, Lester DD, Trainer RJ, Phan T, Kapural L, North JM, Crosby ND, Boggs JW. Percutaneous Peripheral Nerve Stimulation for the Treatment of Chronic Pain Following Amputation. Mil Med. 2019 Jul 1;184(7-8):e267-e274. doi: 10.1093/milmed/usz114. PMID 31111898
- [Background] Ephraim PL, Wegener ST, MacKenzie EJ, Dillingham TR, Pezzin LE. Phantom pain, residual limb pain, and back pain in amputees: results of a national survey. Arch Phys Med Rehabil. 2005 Oct;86(10):1910-9. doi: 10.1016/j.apmr.2005.03.031. PMID 16213230
- [Background] Hanley MA, Ehde DM, Jensen M, Czerniecki J, Smith DG, Robinson LR. Chronic pain associated with upper-limb loss. Am J Phys Med Rehabil. 2009 Sep;88(9):742-51; quiz 752, 779. doi: 10.1097/PHM.0b013e3181b306ec. PMID 19692791
- [Background] Kooijman CM, Dijkstra PU, Geertzen JHB, Elzinga A, van der Schans CP. Phantom pain and phantom sensations in upper limb amputees: an epidemiological study. Pain. 2000 Jul;87(1):33-41. doi: 10.1016/S0304-3959(00)00264-5. PMID 10863043
- [Background] Dijkstra PU, Geertzen JH, Stewart R, van der Schans CP. Phantom pain and risk factors: a multivariate analysis. J Pain Symptom Manage. 2002 Dec;24(6):578-85. doi: 10.1016/s0885-3924(02)00538-9. PMID 12551807
- [Background] Yin Y, Zhang L, Xiao H, Wen CB, Dai YE, Yang G, Zuo YX, Liu J. The pre-amputation pain and the postoperative deafferentation are the risk factors of phantom limb pain: a clinical survey in a sample of Chinese population. BMC Anesthesiol. 2017 May 26;17(1):69. doi: 10.1186/s12871-017-0359-6. PMID 28549447
- [Background] Desmond DM, Maclachlan M. Prevalence and characteristics of phantom limb pain and residual limb pain in the long term after upper limb amputation. Int J Rehabil Res. 2010 Sep;33(3):279-82. doi: 10.1097/MRR.0b013e328336388d. PMID 20101187
- [Background] Schley MT, Wilms P, Toepfner S, Schaller HP, Schmelz M, Konrad CJ, Birbaumer N. Painful and nonpainful phantom and stump sensations in acute traumatic amputees. J Trauma. 2008 Oct;65(4):858-64. doi: 10.1097/TA.0b013e31812eed9e. PMID 18849803
- [Result] Richardson C, Glenn S, Nurmikko T, Horgan M. Incidence of phantom phenomena including phantom limb pain 6 months after major lower limb amputation in patients with peripheral vascular disease. Clin J Pain. 2006 May;22(4):353-8. doi: 10.1097/01.ajp.0000177793.01415.bd. PMID 16691088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One subject was screened and enrolled in this project at a dedicated Pain Center.
Pre-assignment Details: 1 subject was randomized and underwent a crossover treatment.
Groups:
- Treatment Group 2% Lidocaine: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
  First Treatment:
  10 mL 2% lidocaine: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
  Crossover:
  Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
  10 mL preservative free saline: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
- Sham Preservative Free Saline: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
  First Treatment 10 mL preservative free saline: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
  Crossover Treatment 10 mL 2% lidocaine: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
Period: First Intervention
Arm/Group | Treatment Group 2% Lidocaine | Sham Preservative Free Saline
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0
Period: Washout Period 5 Days
Arm/Group | Treatment Group 2% Lidocaine | Sham Preservative Free Saline
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0
Period: Second Intervention (Crossover)
Arm/Group | Treatment Group 2% Lidocaine | Sham Preservative Free Saline
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Project terminated early. PI leaving institution.
Groups:
- Treatment Group 2% Lidocaine: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
  10 mL 2% lidocaine: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
  Crossover: 10 mL preservative free saline: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
- Sham Preservative Free Saline: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
  10 mL preservative free saline: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
  Crossover:10 mL 2% lidocaine: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
- Total: Total of all reporting groups
Arm/Group | Treatment Group 2% Lidocaine | Sham Preservative Free Saline | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: Years] |  | 55 [55 to 55] | 55 [55 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1
Height (Inches) [Mean (Full Range); unit: Inches] |  | 66 [66 to 66] | 66 [66 to 66]
Weight Kilograms [Mean (Full Range); unit: Kilograms] |  | 97 [97 to 97] | 97 [97 to 97]
Level of Amputation [Count of Participants; unit: Participants]
  Above Knee Amputation | 0 | 1 | 1
  Below Knee Amputation | 0 | 0 | 0
Current Pain Level [Mean (Full Range); unit: Score on a scale] — Numeric rating scale (NRS) provided by the participant on a scale of 0 (no pain) to 10 (worst pain imaginable).
  Score on a scale |  | 6 [6 to 6] | 6 [6 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting ≥ 50% Improvement in NRS Pain Score
Description: Proportions of Participants Reporting ≥ 50% Improvement in NRS pain score on a scale of 0 (no pain) to 10 (worst pain imaginable) from baseline at 15 minutes in treatment and sham groups.
Time Frame: 15 minutes after treatment
Population: Only one participant in the trial.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Group 2% Lidocaine: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
  5 days later image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
- Sham Preservative Free Saline: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
  5 Days later:Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
Arm/Group | Treatment Group 2% Lidocaine | Sham Preservative Free Saline
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 24 hours after procedure.
Description: Only one participant was enrolled. The project was closed early due to the investigator leaving the institution.
Groups:
- Treatment Group 2% Lidocaine: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
  10 mL 2% lidocaine: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL 2% lidocaine.
  Crossover:10 mL preservative free saline: Image guided sciatic nerve anesthetic block of the contralateral limb with an injection of 10 mL preservative free saline.
Arm/Group | Treatment Group 2% Lidocaine | Sham Preservative Free Saline
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Study closed early due to PI leaving institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT05046639/Prot_SAP_000.pdf